CLINICAL TRIAL: NCT03740698
Title: The Bio-Inspired Artificial Pancreas for the Home
Acronym: BiAP@home
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17HH3730
Record Dates: First submitted 2018-11-07; First posted 2018-11-14 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a 3-way crossover open-label randomized controlled trial. Description of the three interventions for comparison are as follows:
  1. Sensor augmented pump (combination of insulin pump and continuous glucose monitoring) (open-loop system)
  2. Bio-inspired Artificial Pancreas (closed-loop system) with a fixed bolus calculator
  3. Bio-inspired Artificial Pancreas (closed-loop system) with the Advanced Bolus Calculator for Diabetes (ABC4D)
  The intervention in each arm will be assessed over 6 weeks with a minimum 2-week break in between each intervention. During the break participants will revert back to usual pump therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAP, open-loop (No Intervention): Sensor augmented pump (combination of insulin pump and continuous glucose monitoring) (open-loop system)
- BiAP, fixed bolus calculator (Experimental): Bio-inspired Artificial Pancreas (closed-loop system) with a fixed bolus calculator
  Interventions: Device: BiAP
- BiAP, ABC4D (Experimental): Bio-inspired Artificial Pancreas (closed-loop system) with the Advanced Bolus Calculator for Diabetes (ABC4D)
  Interventions: Device: BiAP; Device: ABC4D

INTERVENTIONS:
Device: BiAP — The bio-inspired artificial pancreas (BiAP) system uses a control algorithm based on a mathematical model of beta-cell behaviour derived from physiological experiments, carried out by other groups, which have demonstrated how the beta cells in the pancreas produce insulin in people without diabetes. Utilising the data from these experiments it has been possible to implement the behaviour of the beta cell in software and we have used a simulator with 200 virtual patients to demonstrate the safety and efficacy of the algorithm. The data from the simulator have previously been published. The BiAP algorithm is implemented on a miniature silicon microchip within a portable handheld device, which interfaces the components of the artificial pancreas.
  Arms: BiAP, ABC4D; BiAP, fixed bolus calculator
Device: ABC4D — The Advanced Bolus Calculator for Diabetes (ABC4D) is a novel, adaptive decision support algorithm based on case-based reasoning (CBR) providing real-time insulin advice through a smartphone application.
  Arms: BiAP, ABC4D

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of a closed-loop insulin delivery system (also known as an artificial pancreas) which is made up of three components that communicate with each other:

1. A glucose sensor that measures glucose every 5 minutes
2. A control algorithm that calculates the required insulin dose
3. An insulin pump that delivers the insulin calculated

DETAILED DESCRIPTION:
In addition to assessing the closed-loop insulin delivery system on its own, the study aims to evaluate the system when combined with a personalised bolus calculator that adapts over time. Standard bolus calculators are widely used in type 1 diabetes self-management to calculate insulin boluses at mealtimes and are incorporated in all insulin pumps and in some glucose meters. A standard bolus calculator uses a generic formula taking into account the target glucose level, current glucose level, carbohydrate content of meal (grams), insulin: carbohydrate ratio (the amount of carbohydrate (grams) covered by 1 unit of insulin), insulin sensitivity factor (the reduction in blood glucose by 1 unit of insulin) and insulin-on-board (IOB, the remaining active insulin from the previous bolus). Some bolus calculators additionally consider parameters such as exercise, but all lack the ability to automatically adapt over time to respond to individual needs.

Finally, the study aims to compare the closed-loop insulin delivery system to standard pump therapy (also known as an open-loop insulin delivery system) in combination with continuous glucose monitoring (referred to as sensor augmented pump).

The Diabetes Technology group at Imperial College have developed a unique closed-loop insulin delivery system known as the Bio-inspired Artificial Pancreas (BiAP) and a personalised bolus calculator known as the Advanced Bolus Calculator for Diabetes (ABC4D).

Overview of the complete closed-loop system (artificial pancreas) used in this study is as follows:

1. A commercially available continuous subcutaneous glucose sensor (Dexcom G5 CGM system).
2. The BiAP control algorithm implemented in a low-power handheld device (developed at Imperial College)
3. An insulin infusion pump (Tandem t:slim) for insulin delivery.

   In one part of the study the closed-loop system will be evaluated in combination with:
4. The ABC4D adaptive bolus calculator implemented in a smartphone (as an app)

All the components will be tested together as a combined system.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Type 1 diabetes confirmed on the basis of clinical features and a random c-peptide <200 pmol/L
* Type 1 diabetes for greater than 1 year
* Continuous subcutaneous insulin infusion for greater than 6 months
* Structured education done (either 1:1 or group education)
* HbA1c <10% (86mmol/mol)
* A negative pregnancy test in female participants of childbearing age

Exclusion Criteria:

* More than one episode of severe hypoglycaemia (defined as hypoglycaemia requiring 3rd party assistance) in the preceding year
* Impaired awareness of hypoglycaemia (Gold score >4)
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Ischaemic heart disease
* Anti-anginal medications
* Regular use of paracetamol
* Unable to participate due to other factors, as assessed by the Chief Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Georgiou P, Toumazou C. A silicon pancreatic Beta cell for diabetes. IEEE Trans Biomed Circuits Syst. 2007 Mar;1(1):39-49. doi: 10.1109/TBCAS.2007.893178. PMID 23851519
- [Background] Oliver N, Georgiou P, Johnston D, Toumazou C. A benchtop closed-loop system controlled by a bio-inspired silicon implementation of the pancreatic beta cell. J Diabetes Sci Technol. 2009 Nov 1;3(6):1419-24. doi: 10.1177/193229680900300623. PMID 20144397
- [Background] Kovatchev BP, Breton M, Man CD, Cobelli C. In silico preclinical trials: a proof of concept in closed-loop control of type 1 diabetes. J Diabetes Sci Technol. 2009 Jan;3(1):44-55. doi: 10.1177/193229680900300106. PMID 19444330
- [Background] Herrero P, Pesl P, Reddy M, Oliver N, Georgiou P, Toumazou C. Advanced Insulin Bolus Advisor Based on Run-To-Run Control and Case-Based Reasoning. IEEE J Biomed Health Inform. 2015 May;19(3):1087-96. doi: 10.1109/JBHI.2014.2331896. PMID 24956470
- [Background] Herrero P, Georgiou P, Oliver N, Johnston DG, Toumazou C. A bio-inspired glucose controller based on pancreatic beta-cell physiology. J Diabetes Sci Technol. 2012 May 1;6(3):606-16. doi: 10.1177/193229681200600316. PMID 22768892

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was put on hold after two participants completed two weeks of the intervention (BIAP) due to technical issues. Due to multiple factors this study has not restarted since and a decision has been made to terminate it.
Period: Overall Study
Arm/Group | SAP, Open-loop | BiAP, Fixed Bolus Calculator | BiAP, ABC4D
Started | 0 | 1 | 1
Completed | 0 | 0 (his study was put on hold after two participants completed two weeks of the intervention (BIAP) due to technical issues. Due to multiple factors this study has not restarted since and a decision has been made to terminate it.) | 0
Not Completed | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Only two of the 8 participants screened and deemed eligible entered an intervention arm. The study was terminate dearly.
Groups:
- Total: Total of all reporting groups
Arm/Group | SAP, Open-loop | BiAP, Fixed Bolus Calculator | BiAP, ABC4D | Total
Number analyzed (Participants) | 0 | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 0 | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: % Time in Target Range Defined as 3.9-10mmol/l
Description: Interstitial blood glucose will be measured every 5 minutes via CGM for a period of six months (original plan)
  The study was terminated early. Only two participants entered the allocated study arm and remained in the study for two weeks.
Time Frame: 6 months
Population: 2 participants with type 1 diabetes. Only two weeks worth of data available for preliminary analysis.
Measure: Number; unit: percentage of time spent in target
Arm/Group | SAP, Open-loop | BiAP, Fixed Bolus Calculator | BiAP, ABC4D
Number analyzed (Participants) | 0 | 1 | 1
percentage of time spent in target |  | 70 | 77

ADVERSE EVENTS:
Time Frame: 2 weeks.
Description: No adverse event.
Arm/Group | SAP, Open-loop | BiAP, Fixed Bolus Calculator | BiAP, ABC4D
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03740698/Prot_SAP_000.pdf